CLINICAL TRIAL: NCT05939804
Title: The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) Application on Patients' Pain Level and Analgesic Use in Patients Undergoing Hip Replacement
Brief Title: The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) Application on Patients' Undergoing Hip Replacement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Acelya Turkmen, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CU-SBF-AT-05
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-07

CONDITIONS: Hip Fractures; Pain, Postoperative; Analgesia
Keywords: Hip Replacement; Transcutaneous Electrical Nerve Stimulation; Pain; Analgesia
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative; Agnosia; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS group (Experimental): 60 minutes of TENS will be applied to the experimental group on the 0th and 1st days after the surgery, and the pain assessment at the time of movement/rest before and after the procedure will be made by the researcher. After the procedure, the amount of analgesic consumed by the experimental group in the first hour will be questioned and recorded.
  Interventions: Device: TENS
- Control group (No Intervention): The routine treatment and care of the control group will not be interfered with.

INTERVENTIONS:
Device: TENS — TENS will be applied to the experimental group on the 0th and 1st days after the surgery, and the pain assessment at the time of movement/rest before and after the procedure will be made by the researcher.
  Arms: TENS group

SUMMARY:
The surgical treatment of an individual with osteoarthritis and hip fracture is provided by hip replacement surgery. While restructuring the joint surfaces with surgery, it is aimed to provide both hip joint movements and to treat pain. Intense perioperative pain after hip replacement is common due to inflammatory agents and surgical intervention (eg, involvement of soft tissue and sensory nerves). Inadequately treated acute postoperative pain causes longer hospital stay, limited and delayed bed rest, decreased compliance with physical therapy, and an increased incidence of postoperative complications. It is thought that this method, which can be effective in the pain control of the patient, will be beneficial for the patient both physiologically and psychologically by reducing pain and discomfort. The most important advantage of TENS; It can be easily applied by nurses and easily taught to patients or families. The nurse has a great role in the follow-up of the patient after the surgery, as she/ he is with the patient for 24 hours. When the literature is examined, it is seen that the number of studies showing the effectiveness of TENS application in patients who underwent hip prosthesis, where studies were conducted with patients with knee gonarthrosis, is limited. In this direction, the aim of the study is to examine the effect of TENS application on patients' pain level and analgesic use in patients undergoing hip replacement.

DETAILED DESCRIPTION:
Intense perioperative pain after hip replacement is common due to inflammatory agents and surgical intervention (eg, involvement of soft tissue and sensory nerves). Inadequately treated acute postoperative pain causes longer hospital stay, limited and delayed bed rest, decreased compliance with physical therapy, and an increased incidence of postoperative complications. Postoperative pain can be treated with narcotics, which is usually accompanied by adverse side effects such as nausea, vomiting, delirium, constipation and gastrointestinal dysfunction. In general, narcotic use should be limited, especially in the elderly, due to the higher incidence of these side effects in this population. However, poor pain management in the elderly not only hinders rehabilitation, but may also lead to other adverse consequences such as tachycardia, increased myocardial oxygen demand, cardiac ischemia and higher risk of post-operative delirium.

Therefore, it is recommended to use non-pharmacological methods as well as pharmacological methods to manage postoperative pain. In the TENS technique, which is one of the non-pharmacological methods used in pain management, a controlled and low-voltage electric current is applied to the nervous system through the skin, and it is seen that the method is used as an effective and non-invasive treatment option in many painful conditions such as neuropathic pain, pain due to osteoarthritis, and post-operative pain. It is thought that this method, which can be effective in the pain control of the patient, will be beneficial for the patient both physiologically and psychologically by reducing pain and discomfort. The most important advantage of TENS; It can be easily applied by nurses and easily taught to patients or families. The nurse has a great role in the follow-up of the patient after the surgery, as she is with the patient for 24 hours. Considering the nursing studies conducted abroad on the application of TENS, it is seen that the nurses apply TENS as a non-pharmacological method in the treatment of pain and train the patients on the application of TENS at home.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* hip replacement insertion
* not have a pacemaker or arrhythmia
* no history of pain, alcohol use or substance abuse
* no history of pain, alcohol use or substance abuse
* no history of pain, alcohol use or substance abuse
* no history of psychiatric illness
* no history of metastatic disease
* being conscious, able to speak
* No barriers to the application of TENS; no postoperative complications
* being I, II and III in the ASA classification of the American Society of Anesthesiology, agreeing to participate in the study.

Exclusion Criteria:

* having a history of epilepsy
* Using analgesics at least 1 hour before TENS is applied
* the presence of a wound in the area where the electrode will be placed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the pain level using the VAS. | 48 hour
  Reducing the pain level of patients undergoing hip replacement by applying TENS.
  A value of 0 on the scale means that the patient does not experience pain, and a value of 10 means that he experiences pain at the most severe level
Change in analgesic consumption | 48 hour
  Changing analgesic consumption of patients by applying TENS. The analgesic consumption in the first 2 days after the surgery will be learned by using the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Açelya Türkmen, PhD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No